CLINICAL TRIAL: NCT00902278
Title: Immune Response Induced by Different Manufacturers of Influenza Vaccines
Brief Title: Immune Responses Induced by Different Licensed Influenza Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Mary Co, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H 13000
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-06

CONDITIONS: Immune Response
Keywords: influenzavirus A; influenzavirus B; human influenza; T lymphocytes; influenza vaccines
MeSH Terms: conditions — Influenza, Human | interventions — FluLaval; Influenza Vaccines; fluarix; Afluria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Flulaval (Active Comparator)
  Interventions: Biological: Flulaval
- Fluvirin (Active Comparator)
  Interventions: Biological: Fluvirin
- Fluzone (Active Comparator)
  Interventions: Biological: Fluzone
- Fluarix (Active Comparator)
  Interventions: Biological: Fluarix
- Affluria (Active Comparator)
  Interventions: Biological: Afluria

INTERVENTIONS:
Biological: Flulaval — one 0.5-mL dose via intramuscular injection
  Arms: Flulaval
Biological: Fluvirin — one 0.5-mL dose via intramuscular injection
  Arms: Fluvirin
Biological: Fluzone — one 0.5-mL dose via intramuscular injection
  Arms: Fluzone
Biological: Fluarix — one 0.5-mL dose via intramuscular injection
  Arms: Fluarix
Biological: Afluria — one 0.5-mL dose via intramuscular injection
  Arms: Affluria

SUMMARY:
The goal of this research is to find out how the body's immune system responds to different manufacturer's "flu" vaccines.

DETAILED DESCRIPTION:
There are currently five licensed inactivated influenza vaccines approved for use in the United States by the Food and Drug Administration.Current influenza virus vaccines consist of 3 components: the HA protein from an H1N1 virus, an H3N2 and an influenza B virus.Influenza vaccines are evaluated and approved by the FDA on the basis of HA and NA content. However, different manufacturing processes are involved in the preparation of these commercial vaccines and evidence suggests that each of these vaccines contain similar patterns of HA protein but different patterns of influenza influenza internal proteins such as NP and M1. The presence of these additional internal proteins of influenza virus which are targets of T cell responses suggest not only the potential for additional protection derived from influenza vaccines other than antibody mediated protection but also differential levels of T cell mediated protection between different manufacturers of commercial influenza vaccines.Each subject will have four blood samples taken- prevaccination and at Days 7, 14,30 and 3-5 months post vaccination. These samples will be tested for T and B cell responses and the results compared between different manufacturers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-50 years of age)
* Willing to donate a blood sample multiple times
* Willing to sign informed consent and HIPAA

Exclusion Criteria:

* Known systemic hypersensitivity reactions to egg proteins (eggs or egg products), to chicken proteins
* Known hypersensitivity to neomycin, thimerosol (mercury derivative), neomycin, or polymyxin
* Previous life threatening reaction to influenza vaccine
* Individuals with altered immunocompetence state from medical condition ( HIV, cancer) or through immunosuppressive therapy(irradiation,corticosteroids, antimetabolites, alkylating agents, cytotoxic agents)
* Occurrence of neurological syndrome within six weeks of previous influenza immunization
* Active neurological disorder characterized by changing neurological disorder
* Pregnancy
* Acute febrile illness
* History of anemia or bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2008-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dawn T Co, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited healthy adults subjects during the 2008-2009, 2009-2010, 2010-2011, and 2011-2012 influenza seasons in a clinical research setting.
Period: Overall Study
Arm/Group | Flulaval | Fluvirin | Fluzone | Fluarix | Afluria
Started | 54 | 36 | 54 | 12 | 37
Completed | 50 | 34 | 49 | 12 | 35
Not Completed | 4 | 2 | 5 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 3 | 2 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flulaval | Fluvirin | Fluzone | Fluarix | Afluria | Total
Number analyzed (Participants) | 54 | 36 | 54 | 12 | 37 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 36 | 54 | 12 | 37 | 193
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 32 | 37 | 6 | 25 | 141
  Male | 13 | 4 | 17 | 6 | 12 | 52
Region of Enrollment [Number; unit: participants]
  United States | 54 | 36 | 54 | 12 | 37 | 193

OUTCOME MEASURES:

1. Primary Outcome: T Cell Responses Following Immunization
Description: Comparison of mean peak fold increases in ELISPOT H1N1, H3N2, and B responses between different vaccine groups
Time Frame: Prevaccination and approximately 7 days,14 days ,1month and up to 3-5 months post vaccination
Population: Data was collected only for participants from the 2008-2009 influenza season. Data was not collected for Flulaval group.Only participants with evaluable data were included in the analysis.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Flulaval | Fluvirin | Fluzone | Fluarix | Afluria
Number analyzed (Participants) | 0 | 10 | 12 | 11 | 12
fold change
  H1N1 virus |  | 1.5 (.55) | 1.7 (.84) | 1.9 (.56) | 1.6 (.71)
  H3N2 virus |  | 2.4 (1.28) | 2.1 (1.34) | 2.7 (1.23) | 1.7 (.60)
  B virus |  | 1.5 (.61) | 1.6 (.59) | 1.6 (.59) | 1.4 (.61)

2. Secondary Outcome: Antibody Responses Following Immunization
Description: Geometric mean fold rise in antibody titer between day 0 ( baseline) and approximately 1 month post vaccination within each vaccine group
Time Frame: Prevaccination and approximately 1 month post vaccination
Population: Data was collected only for participants from the 2008-2009 influenza season. Data was not collected for the flulaval group. Only participants with evaluable data were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Flulaval | Fluvirin | Fluzone | Fluarix | Afluria
Number analyzed (Participants) | 0 | 11 | 12 | 12 | 12
fold change
  H1N1 |  | 7.32 [-61.28 to 75.92] | 7.02 [-54.6 to 68.62] | 5.71 [-9.49 to 20.91] | 5.26 [-5.88 to 16.4]
  H3N2 |  | 7.6 [-30.1 to 45.3] | 7.2 [-74.8 to 89.2] | 4.9 [-6.2 to 16] | 5.6 [-14.9 to 26.1]
  B |  | 3.4 [-41.6 to 48.4] | 9.3 [-34 to 52.6] | 9.6 [-52.99 to 72.21] | 4.0 [-6.9 to 14.9]

ADVERSE EVENTS:
Description: Only participants with available data were included in the analysis.
Arm/Group | Flulaval | Fluvirin | Fluzone | Fluarix | Afluria
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/34 | 0/53 | 0/11 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/34 | 0/53 | 0/11 | 0/36
Other Adverse Events (participants affected / at risk) | 30/52 | 24/34 | 32/53 | 6/11 | 25/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flulaval (N=52) | Fluvirin (N=34) | Fluzone (N=53) | Fluarix (N=11) | Afluria (N=36)
Headache (Nervous system disorders) | 8 (8) | 6 (6) | 8 (8) | 4 | 4 (4)
Injection site soreness/tenderness (Skin and subcutaneous tissue disorders) | 17 (17) | 10 (10) | 11 (11) | 1 (1) | 13 (13)
Arm soreness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 | 9 (9) | 1 (1) | 8 (8) — Soreness or tenderness
Sore throat (Gastrointestinal disorders) | 4 (4) | 6 (6) | 4 (4) | 0 | 4 (4) — Scratchy or sore throat
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3) | 0 | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 0 | 3 (3)
Fatigue (General disorders) | 3 (3) | 4 (4) | 4 (4) | 0 | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 | 0 (0) | 1 | 0 (0) — Includes neck, back, shoulder pain
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 | 0 (0)
Sniffles (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 | 0 (0)
Muscle stiffness/achiness/pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4) | 1 | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 | 0 (0) — abdominal pain or cramps
" Cold symptoms" (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 3 (3) | 0 | 1 (1)
fevers (Infections and infestations) | 2 (2) | 0 | 1 | 1 | 3 (3) — fevers, feverish,
nausea (Gastrointestinal disorders) | 1 (1) | 1 | 2 (2) | 1 | 2 (2)
injection site swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 | 1 | 1 | 0
sweats (Metabolism and nutrition disorders) | 0 (0) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No